CLINICAL TRIAL: NCT02838849
Title: Fiber and Water Improve Bowel Habit and Stool Microbiota in Healthy Participants: a Randomized Clinical Trial
Brief Title: Fiber and Water Improve Bowel Habit in Humans
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universidade de Passo Fundo (Other)
Responsible Party: Principal Investigator, Fernando Fornari, Professor, Universidade de Passo Fundo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MASTERUFRGSGROSA
Record Dates: First submitted 2016-07-11; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Dietary Habits; Bowel Dysfunction
MeSH Terms: conditions — Feeding Behavior; Intestinal Diseases | interventions — Dietary Fiber; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fiber (Sham Comparator): Participants were treated with 2 sachets of fiber orally a day for 14 days, after baseline characterization of bowel habit and stool features.
  Interventions: Dietary Supplement: Fiber
- Fiber and Water (Active Comparator): Participants were treated with 2 sachets of fiber orally a day and ingested 2 liters of water a day for 14 days, after baseline characterization of bowel habit and stool features.
  Interventions: Dietary Supplement: Fiber and Water

INTERVENTIONS:
Dietary Supplement: Fiber — Fiber composed of wheat bran, pectin and green banana flour (total daily amount of 13 g for women and 20 g for men), keeping the usual liquid intake
  Arms: Fiber
Dietary Supplement: Fiber and Water — Fiber composed of wheat bran, pectin and green banana flour (total daily amount of 13 g for women and 20 g for men) plus 2 liter of water/day
  Arms: Fiber and Water

SUMMARY:
Twenty healthy volunteers had their baseline parameters (symptoms, bowel habit, quality of life, fecal characteristics and microbiota) measured during a week of monitoring followed by randomization to a 14 days course of increased fiber in diet or increased fiber and water intake, with repetition of parameters measuring at the end.

DETAILED DESCRIPTION:
Demographic and clinical data were collected and recorded in the first interview after signing the informed consent. The protocol was composed of two phases. The baseline phase lasted 7 days, when participants reported their usual diet on a food dairy in the first 3 days, between Sunday and Tuesday. Calculation of nutrient intake was performed using ADS nutri software (UFPEL, Pelotas, Brazil). Participants approved for the next phase were then randomized to fiber and fiber+water groups, which lasted 14 days. During this period participants were asked to report their intestinal habits including bowel movements, graduation of straining and subjective stool consistency. Participants were instructed to rank straining using a Likert scale from 1 (minimum) to 5 (maximum), and the Bristol scale for stool consistency. In the last day of treatment phase (Saturday) participants collected feces and urine of 24 hours, and responded a symptoms questionnaire. Food and liquid intake were recorded on a diary during the last 3 days of treatment for comparison with the baseline phase stage.

ELIGIBILITY:
Inclusion Criteria:

* non-obese
* absence of abdominal complaints

Exclusion Criteria:

* use of medications that interfere with the gastrointestinal tract function
* past of abdominal surgery
* any acute or chronic disease

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
bowel habit: evacuation frequency | 14 days
  The patient reported in a diary the number of evacuations per day during 14 days of experimental use of fiber or fiber+water
bowel habit: straining | 14 days
  The patient reported the effort for each evacuation using a Likert scale between 1 and 5 (1 = no effort / 5 = maximal) during 14 days of experimental use of fiber or fiber+water
bowel habit: stool consistency | 14 days
  The patient reported the stool consistency of evacuations using a Bristol scale during 14 days of experimental use of fiber or fiber+water

SECONDARY OUTCOMES:
Abdominal symptoms | 14 days
  self report of any abdominal symptom (yes/not) during treatment with fiber or fiber+water, including: pain, discomfort, distension, defecation urgency, backpain
Stool characteristics: fecal weight | 14 days
  A sample of feces was collected at the end of 14 days treatment and analyzed for fecal weight (g)
Stool characteristics: percentage of water | 14 days
  A sample of feces was collected at the end of 14 days treatment and analyzed for water percentage
Stool characteristics: pH | 14 days
  A sample of feces was collected at the end of 14 days treatment and analyzed for measurement of pH
Intestinal microbiota | 14 days
  A sample of feces was collected at the end of 14 days treatment for PCR analyses of 10 bacteria groups.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Fornari, Professor, Principal Investigator — Universidade de Passo Fundo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goncalves GVR, Canova R, Callegari-Jacques SM, Frandoloso R, Kreutz LC, Fornari F. Short-term intestinal effects of water intake in fibre supplementation in healthy, low-habitual fibre consumers: a phase 2 clinical trial. Int J Food Sci Nutr. 2022 Sep;73(6):841-849. doi: 10.1080/09637486.2022.2079117. Epub 2022 May 23. PMID 35603590